CLINICAL TRIAL: NCT06050096
Title: Drug-coated Balloons Treatment in Chronic Total Occlusion Coronary Artery Disease Guided by Intravascular Ultrasound
Brief Title: DCB Treatment in CTO Guided by IVUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Principal Investigator, Chenpengsheng, principal investigator, Xuzhou Central Hospital
Other Study IDs: 001
Record Dates: First submitted 2023-09-08; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DCB group: CTO patients treated by DCB
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — CTO patients treated by DCB

SUMMARY:
The percutaneous coronary intervention (PCI) for chronic total occlusion (CTO) coronary artery disease is difficult, the success rate is low, and the incidence of re-occlusion and restenosis is high. With the wide application of imaging technology represented by intravascular ultrasound (IVUS), the success rate of CTO PCI has been significantly improved. Drug-coated balloons (DCB), as a treatment without metal implantation, has lower lumen loss and no significant increase in the rate of revascularization. Through IVUS measurement of vascular lumen after CTO opening, appropriate instruments can be selected for adequate dilation, and appropriate treatment methods can be selected according to different lumen structures. Therefore, the purpose of this study was to evaluate the clinical effect of IVUS-guided DCB therapy on CTO lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18, male or female;
2. Patients who meet the diagnostic criteria for coronary heart disease, have clinical symptoms and seek interventional treatment;
3. Coronary angiography confirmed that the blood vessels met the diagnostic criteria of CTO;
4. Sign informed consent and be willing to undergo follow-up for at least 12 months.

Exclusion Criteria:

1. Patients with severe contrast allergy who cannot tolerate coronary angiography;
2. Patients known allergy to drug balloon coating;
3. Patients who is pregnant or breastfeeding;
4. Bleeding or other diseases, such as digestive tract ulcers, blood system diseases, etc., limit the use of platelet aggregation inhibitors and anticoagulation therapy;
5. Patients with cardiac shock;
6. Patients with a life expectancy of less than 1 year;
7. Other situations deemed unsuitable for inclusion by the researcher.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Among CTO lesions previously treated with DCB, the incidence of restenosis was 11.8%, with a sample size of 90-110. This is an observational study on the treatment of CTO, and all patients with CTO lesions were nonselectively enrolled. Continuous enrollment of CTO patients from September 2023 to August 2024 (an estimated 100 cases) was designed to observe the clinical effect of IVUS-directed DCB therapy on CTO lesions.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of major adverse cardiovascular events (MACE) in 12 month | 12 month
  cardiovascular death, nonfatal myocardial infarction, and target vessel revascularization

SECONDARY OUTCOMES:
Rate of cardiovascular death in 12 month | 12 month
Rate of nonfatal myocardial infarction in 12 month | 12 month
Rate of target vessel revascularization in 12 month | 12 month
Rate of procedure success rate after PCI | 1 day
Rate of technical success after PCI | 1 day
Rate of minor bleeding events | 12 month
Rate of major bleeding events | 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Result] Tajti P, Burke MN, Karmpaliotis D, Alaswad K, Werner GS, Azzalini L, Carlino M, Patel M, Mashayekhi K, Egred M, Krestyaninov O, Khelimskii D, Nicholson WJ, Ungi I, Galassi AR, Banerjee S, Brilakis ES. Update in the Percutaneous Management of Coronary Chronic Total Occlusions. JACC Cardiovasc Interv. 2018 Apr 9;11(7):615-625. doi: 10.1016/j.jcin.2017.10.052. Epub 2018 Mar 14. PMID 29550088
- [Result] Di Mario C, Werner GS, Sianos G, Galassi AR, Buttner J, Dudek D, Chevalier B, Lefevre T, Schofer J, Koolen J, Sievert H, Reimers B, Fajadet J, Colombo A, Gershlick A, Serruys PW, Reifart N. European perspective in the recanalisation of Chronic Total Occlusions (CTO): consensus document from the EuroCTO Club. EuroIntervention. 2007 May;3(1):30-43. No abstract available. PMID 19737682
- [Result] Werner GS, Gitt AK, Zeymer U, Juenger C, Towae F, Wienbergen H, Senges J. Chronic total coronary occlusions in patients with stable angina pectoris: impact on therapy and outcome in present day clinical practice. Clin Res Cardiol. 2009 Jul;98(7):435-41. doi: 10.1007/s00392-009-0013-5. Epub 2009 Mar 18. PMID 19294443
- [Result] Brilakis ES, Karmpaliotis D, Patel V, Banerjee S. Complications of Chronic Total Occlusion Angioplasty. Interv Cardiol Clin. 2012 Jul;1(3):373-389. doi: 10.1016/j.iccl.2012.04.006. Epub 2012 May 31. PMID 28582023
- [Result] Madhavan MV, Kirtane AJ, Redfors B, Genereux P, Ben-Yehuda O, Palmerini T, Benedetto U, Biondi-Zoccai G, Smits PC, von Birgelen C, Mehran R, McAndrew T, Serruys PW, Leon MB, Pocock SJ, Stone GW. Stent-Related Adverse Events >1 Year After Percutaneous Coronary Intervention. J Am Coll Cardiol. 2020 Feb 18;75(6):590-604. doi: 10.1016/j.jacc.2019.11.058. PMID 32057373
- [Result] Kereiakes DJ. The TWENTE Trial in Perspective: Stents and Stent Trials in Evolution. JAMA Cardiol. 2017 Mar 1;2(3):235-237. doi: 10.1001/jamacardio.2016.5208. No abstract available. PMID 28114677
- [Result] Buccheri D, Lombardo RM, Cortese B. Drug-coated balloons for coronary artery disease: current concepts and controversies. Future Cardiol. 2019 Nov;15(6):437-454. doi: 10.2217/fca-2019-0009. Epub 2019 Nov 5. PMID 31686536
- [Result] Giacoppo D, Alfonso F, Xu B, Claessen BEPM, Adriaenssens T, Jensen C, Perez-Vizcayno MJ, Kang DY, Degenhardt R, Pleva L, Baan J, Cuesta J, Park DW, Kukla P, Jimenez-Quevedo P, Unverdorben M, Gao R, Naber CK, Park SJ, Henriques JPS, Kastrati A, Byrne RA. Drug-Coated Balloon Angioplasty Versus Drug-Eluting Stent Implantation in Patients With Coronary Stent Restenosis. J Am Coll Cardiol. 2020 Jun 2;75(21):2664-2678. doi: 10.1016/j.jacc.2020.04.006. PMID 32466881
- [Result] Koln PJ, Scheller B, Liew HB, Rissanen TT, Ahmad WA, Weser R, Hauschild T, Nuruddin AA, Clever YP, Ho HH, Kleber FX. Treatment of chronic total occlusions in native coronary arteries by drug-coated balloons without stenting - A feasibility and safety study. Int J Cardiol. 2016 Dec 15;225:262-267. doi: 10.1016/j.ijcard.2016.09.105. Epub 2016 Sep 27. PMID 27741486
- [Result] Jeger RV, Eccleshall S, Wan Ahmad WA, Ge J, Poerner TC, Shin ES, Alfonso F, Latib A, Ong PJ, Rissanen TT, Saucedo J, Scheller B, Kleber FX; International DCB Consensus Group. Drug-Coated Balloons for Coronary Artery Disease: Third Report of the International DCB Consensus Group. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1391-1402. doi: 10.1016/j.jcin.2020.02.043. Epub 2020 May 27. PMID 32473887
- [Result] Wohrle J, Zadura M, Mobius-Winkler S, Leschke M, Opitz C, Ahmed W, Barragan P, Simon JP, Cassel G, Scheller B. SeQuentPlease World Wide Registry: clinical results of SeQuent please paclitaxel-coated balloon angioplasty in a large-scale, prospective registry study. J Am Coll Cardiol. 2012 Oct 30;60(18):1733-8. doi: 10.1016/j.jacc.2012.07.040. Epub 2012 Oct 3. PMID 23040575
- [Result] Jun EJ, Shin ES, Teoh EV, Bhak Y, Yuan SL, Chu CM, Garg S, Liew HB. Clinical Outcomes of Drug-Coated Balloon Treatment After Successful Revascularization of de novo Chronic Total Occlusions. Front Cardiovasc Med. 2022 Apr 13;9:821380. doi: 10.3389/fcvm.2022.821380. eCollection 2022. PMID 35498010
- [Result] Yuan SL, Kim MH, Garg S, Shin ES. A case of drug-coated balloon treatment for two total occluded lesions in a patient with acute coronary syndrome. Cardiol J. 2020;27(3):320-321. doi: 10.5603/CJ.2020.0083. No abstract available. PMID 32583405
- [Result] Huang WC, Teng HI, Hsueh CH, Lin SJ, Chan WL, Lu TM. Intravascular ultrasound guided wiring re-entry technique for complex chronic total occlusions. J Interv Cardiol. 2018 Oct;31(5):572-579. doi: 10.1111/joic.12518. Epub 2018 May 3. PMID 29726047